CLINICAL TRIAL: NCT07028385
Title: Exploratory Phase 2 Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Safety and Impact on HIV-1 Reservoir of Baricitinib in Virologically Suppressed People With HIV-1
Brief Title: Safety and Impact of Baricitinib on Cell Surivival Pathways, HIV-1 Reservoir and Inflamation in People With HIV-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: IrsiCaixa (Other); University of Turin, Italy (Other); Instituto de Salud Carlos III (Other Government); Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCN05-Bari; 2024-520159-26-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-10

CONDITIONS: HIV
Keywords: bariticinib; HIV; ctl resistance; jak/stat inhibitor; bcl2

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 2:1 to the 2 arms: Bariticinib arm VS Placebo arm
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Bariticinib will be re-encapsulated with identical weight and appearance (shape, size, colour and flavour) as the placebo-containing capsules.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bariticinib (Experimental): Participants will take one capsule containing 2 mg of baricitinib, once daily, oral administration for 12 weeks
  Interventions: Drug: Bariticinib 2 mg
- Placebo (Placebo Comparator): Participants will take one capsule containing inert substance (maltodextrine), once daily, oral administration for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bariticinib 2 mg — Commercially available tablets containing 2 mg of barticiinib will be used. The tablets will be re-capsulated to keep the study blind.
  Arms: Bariticinib
Other: Placebo — Maltodextrin capsules with identical weight and appearance (shape, size, colour and flavour) as the bariticinib-containing capsules.
  Arms: Placebo

SUMMARY:
The goal of this exploratory clinical trial is to evaluate the safety and tolerability of bariticinib administered at 2 mg once daily during 12 weeks in 30 people living with HIV-1 (PWH) on suppressive antiretroviral therapy (ART) and to evaluate changes in levels of phosphorylated STAT (pSTAT) after 12 weeks of treatment with bariticinib. The main questions it aims to answer are:

* The safety and tolerability of bariticinib
* To evaluate the effects of bariticinib on T-cells (HIV-1 reservoirs, apoptosis, inflamation, activation and exhaustion).
* To characterize bariticinib pharmacokinetics in plasma.

Participants will be treated with pral Barticinib 2mg or matched Placebo daily for 12 weeks. Suppressive cART will remain unchanged during the entire study. Participants will be followed until week 24, in a total of 8 visits.

DETAILED DESCRIPTION:
Despite the success of antiretroviral therapy (ART) in suppressing HIV replication, it does not eliminate the latent viral reservoir, which remains a major barrier to achieving a cure. Recent evidence suggests that HIV-infected cells may evade immune clearance by overexpressing anti-apoptotic proteins such as BCL-2, contributing to reservoir persistence. Baricitinib, a second-generation Janus kinase (JAK) inhibitor has shown potential in preclinical studies to reduce HIV reactivation and modulate immune activation.

This study investigates whether baricitinib can safely modulate the HIV-1 reservoir and immune environment in PWH on suppressive ART.

Participants will be randomized (2:1) to receive either oral baricitinib 2 mg or placebo daily for 12 weeks, followed by a 12-week observation period.

The primary objectives are to assess the safety and tolerability of baricitinib and to evaluate changes in phosphorylated STAT (pSTAT) levels in CD4+ T cells as a pharmacodynamic marker.

Secondary objectives include evaluating the effects of baricitinib on BCL-2 expression, JAK/STAT signaling, HIV-1 reservoir size, inflammatory biomarkers, and immune cell subsets.

Exploratory analyses will assess HIV-specific T cell responses, CD4+ T cell susceptibility to cytotoxic T lymphocyte (CTL) killing, and transcriptomic changes.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged between 18 and 65 years on the day of screening visit.
* Confirmed HIV-1 infection.
* Receiving suppressive cART for at least 2 years (defined as maintained plasma viral load <50 copies/mL, allowing for isolated blips [<200 cop/ml, non-consecutive, representing <20% total determinations]).
* Being on the same cART regimen within at least 4 weeks prior to baseline visit (week 0).
* Willing and able to be adherent to their cART regimen for the duration of the study.
* Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study.
* In the opinion of the clinical Investigator, the candidate has understood the information provided and can give written Informed Consent.
* If heterosexually active female of childbearing potential using an effective method of contraception different from hormonal contraception (intra-uterine device (IUD), anatomical sterility in self or partner or sexual abstinence) from 14 days prior to the first IMP administration and commit to use it until 3 months after the last IMP administration. All female candidates of childbearing potential who are not sexually active with men at screening, must agree to utilize an effective method of contraception if they become sexually active during the study.
* If female of childbearing potential, willing to undergo urine pregnancy tests at the designated time points.
* If positive IgG for varicella zoster, adequate herpes zoster vaccination at least 4 weeks prior to week 0 visit.
* Willing to accept blood draws at time points specified in the Schedule of Events.

Exclusion Criteria:

* If female of childbearing potential, pregnant or planning a pregnancy during the entire study or lactating.
* Prior history or clinical manifestations of any physical or psychiatric disorder that could impair the subject's ability to complete the study.
* Any active AIDS-defining disease or progression of HIV-related disease, except cutaneous Kaposi's sarcoma not requiring systemic therapy.
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical, anal, or penile intraepithelial neoplasia.
* Systemic treatment for cancer within 1 year of study entry.
* Known hypersensitivity to any component of the IMP formulation, or severe or multiple allergies to drugs or pharmaceutical agents.
* Potential participant received or plans to receive:

  i. Licensed live attenuated vaccines within 28 days before or after inflammation and immune biomarkers visit (weeks 0 and 12).

ii. Other vaccines (eg, tetanus, hepatitis A, hepatitis B, rabies, pneumococcal, recombinant Herpes Zoster, Influenza, COVID-19 vaccines) within 14 days before or after inflammation and immune biomarkers visits (weeks 0 and 12).

* Receipt of blood products within 3 months of study entry.
* Current or recent use (within last 3 months) of interferon or systemic corticosteroids or other immunosuppressive agents (use on inhaled steroids for asthma or topic steroids for localized skin conditions are permitted).
* Any other current or prior therapy which, in the opinion of the investigator, would make the individual unsuitable for the study or influence the results of the study.
* Prior history of thrombotic events (deep venous thrombosis, pulmonary embolism, or arterial thrombosis) or known inherited prothrombotic disorders (Factor V Leiden, prothrombin G2021A mutation, antithrombin deficiency, protein S deficiency, protein C deficiency, etc).
* Current use of combined hormonal contraceptives or substitutive hormonal treatment.
* History of any of the following cardiovascular diseases: myocardial infarction, unstable angina, congestive heart failure, uncontrolled arrhythmias, cardiac revascularization, stroke, uncontrolled hypertension, or uncontrolled diabetes within 6 months.
* Current smokers over 10 cigarettes per day or former smokers with a history of smoking more than 10 packyears, unless they quit smoking more than 15 years ago.
* Positive hepatitis C IgG, unless confirmed clearance of HCV infection (undetectable plasma viral load, spontaneous or following treatment).
* Chronic hepatitis B, defined as positive hepatitis B surface antigen (HBsAg); or past hepatitis B, defined as positive hepatitis B core antibody (HBcAb), unless ART regimen contains FTC/TFV during the study.
* Symptomatic herpes zoster or recurrent genital herpes within 24 weeks, or any history of disseminated herpes simplex, disseminated herpes zoster, ophthalmic zoster, or CNS zoster.
* History of active, past, or latent tuberculosis, confirmed through medical history, clinical records, or a positive TB IGRAs by QuantiFERON test, unless documented preventive TB treatment with 6 or 9 months of daily isoniazid, or a 3-month regimen of weekly rifapentine plus isoniazid, or a 3-month regimen of daily isoniazid plus rifampicin.
* Any laboratory abnormalities including:

Hematology

* Hemoglobin <10.0 g/dl,
* Absolute neutrophil count ≤1,000 /mm3,
* Absolute lymphocyte count ≤500 /mm3,
* Platelets >450,000/mm3, Biochemistry
* eGFR <30 ml/min,
* AST > 2.5 x ULN,
* ALT > 2.5 x ULN,

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of baricitinib. | From baseline (week 0) to week 12
  Proportion of participants developing Grade 3 or 4 treatment-related adverse events or laboratory abnormalities during the study, based on the Division of AIDS (DAIDS) Table for grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 [July 2017].
To evaluate changes in levels of phosphorylated STAT (pSTAT) in CD4+ T cells, as a pharmacodynamic biomarker of baricitinib activity. | From baseline (week 0) to week 12
  Levels of pSTAT 1, 3 and 5 in CD4+ T cells measured by Flow cytometry.

SECONDARY OUTCOMES:
To evaluate the effect of baricitinib on proapoptotic pathways mediated by BCL-2. | From baseline (week 0) to week 12
  Changes in levels of BCL-2 in CD4+ T cells measured by Flow cytometry.
To evaluate the effect of baricitinib on JAK/STAT signaling pathway | From baseline (week 0) to week 12
  Changes in levels of IFITM2, pJAK1/2, cleaved-caspase 3 and other proapoptotic markers in CD4+ T cells measured by Western blot.
To evaluate the effect of baricitinib on the HIV-1 reservoir. | From baseline (week 0) to week 12
  Changes in total and intact proviral HIV-1 DNA (IPDA) in CD4 T cells.
To evaluate the impact of baricitinib on homeostatic cytokines, inflammatory biomarkers and cell death markers. | From baseline (week 0) to week 12
  Changes in soluble plasma levels of proinflammatory biomarkers (such as IL-2, IL-6, IL-7, IL-15, IL-8, TNFa, IFNg and sCD14) and anti-inflammatory biomarkers (such as IL-10, IL-4, IL-13).
To evaluate the effects of baricitinib in immune cell subsets. | From baseline (week 0) to week 12
  Changes in T cell immune subsets and frequencies of T cells expressing activation, exhaustion and senescence markers measured by multiparametric flow cytometry.
To characterize baricitinib pharmacokinetics in plasma. | From week 4 to week 12
  Baricitinib concentrations in plasma

OTHER OUTCOMES:
To evaluate the effect of baricitinib in HIV-1 specific T cells. | From baseline (week 0) to week 12
  Changes in HIV-specific CD8 T cells responses measured by AIM/ICS flow cytometry after peptide stimulation, IFNg ELISPOT, proliferation and/or viral suppressive assays.
To evaluate the effect of baricitinib on CD4 sensitivity to CTL killing. | From baseline (week 0) to week 12
  Changes in surviving CD4 T cells using peptide-pulsed isolated CD4 T cells co-cultured with autologous CD8.
To assess the impact of baricitinib on transcriptomic signatures related to survival, apoptotic regulation (both pro- and anti-apoptotic), and activation pathways. | From baseline (week 0) to week 12
  Changes in gene expression profiles focused on cell death, apoptosis and viral transcription factors by RNAseq in isolated CD4+ and CD8+ T cells

CONTACTS AND LOCATIONS:
Locations (1):
- Fundació Lluita contra les Infeccions - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared publicly due to the exploratory nature of the trial, the limited sample size, and the sensitive nature of the data related to HIV status and immunological profiling.